CLINICAL TRIAL: NCT05236595
Title: Research for Individualized Therapeutics in Rare Genetic Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Margot A. Cousin, Principal Investigator, Mayo Clinic
Other Study IDs: 21-006562
Record Dates: First submitted 2021-12-27; First posted 2022-02-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Rare Genetic Disease; Undiagnosed Diseases
MeSH Terms: conditions — Undiagnosed Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Research blood collection kits will attempt to be collected on all active study participants. Other biospecimens including fibroblasts, CSF, saliva, buccal swabs, and tissue may also be collected under the protocol as needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rare genetic disease individualized drug development screening candidate: Patients with targetable disease-causing genetic alterations will be evaluated on a case by case basis. The research study will utilize biospecimens to determine if an individualized therapeutic may be developed as a possible treatment option. If an individualized therapeutic drug can be developed, a future IND FDA application (n=1) will be filed.
  Interventions: Other: Individualized drug matching per genetic disease

INTERVENTIONS:
Other: Individualized drug matching per genetic disease — Patient phenotype and samples will be evaluated for individualized therapeutic drug development

SUMMARY:
The purpose of this research study is to identify individuals that have a rare genetic disease without an adequate therapeutic strategy that might be treatable with drug developed to target the disease-causing genetic alteration.

ELIGIBILITY:
Inclusion Criteria:

* Has Mayo Clinic or other medical health system ID, or another unique identifier.
* Able to provide informed consent.
* Individual must have evidence of a genetic disorder as determined by a provider or genetic counselor with causative or likely causative genetic variants identified by molecular testing.
* Genetic variants must be hypothesized to be targetable using antisense oligonucleotide drugs (such as: knockdown gain of function alterations, increase protein production for reduced function alterations, or modulate mRNA splicing to correct abnormal splicing, promote normal splicing, or return reading frame to an out-of-frame transcript to restore function, etc.) based on current acceptable understanding of ASO mechanisms of action and tissue/organ targeting efficiency.
* Biological family member of an enrolled individual.
* Would be able to travel to a Mayo Clinic site for ongoing treatment should a therapeutic be developed.
* Treatment at the individual's current disease state would likely provide benefit based on current clinical data and understanding of the progression of the disease.

-Or-

* Biological family member of an enrolled individual
* Able to provide informed consent or has a LAR available to provide informed consent

Exclusion Criteria

* Individuals who have situations that would limit compliance with the study requirements.
* Institutionalized (i.e. Federal Medical Prison).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have been diagnosed with a rare genetic disorder for which adequate or curative treatment is not currently available.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Enrollment of study participants | 5 years
  To recruit and enroll participants with a confirmed rare genetic disease whose genetic variants may be targetable by an ASO and/or other drug.
Collection of biospecimens | 5 years
  Total number of biopecimens collected which may include blood samples, skin biopsy and fibroblast culture, organ biopsy specimens
Partnered research with external entities | 5 years
  To engage in partnered research with external entities (foundations, academia, and drug companies) to facilitate the ASO and/or other drug development and testing.
Future IND applications | 5 years
  To submit an IND application with the FDA following successful drug development and safety/toxicity testing outcomes.
Determine natural history and clinical baseline | 5 years
  To determine the natural history and clinical baseline of patient's disease status. This will be used to determine efficacy when treated with experimental ASO and/or other drug.
Determine individualized therapeutic efficacy | 5 years
  To determine clinical efficacy of treatment with experimental ASO and/or other drug.
Publish findings | 5 years
  To publish and/or share findings to improve patient specific ASO and/or other drug development and increase the number of therapeutic options for individuals with rare genetic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Margot A Cousin, Ph.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Minneota, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials